CLINICAL TRIAL: NCT00687596
Title: A Phase 2, Double-blind, Placebo-controlled, Randomized, International, Multicenter Study of Oral TAC 101 as Second Line Treatment in Patients With Advanced Hepatocellular Carcinoma Who Received Sorafenib as First Line Therapy
Brief Title: Study of TAC-101 as Second Line Treatment in Patients With Advanced Hepatocellular Carcinoma Who Received Sorafenib as First Line Therapy
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Terminated due to safety concerns
Sponsor: Taiho Oncology, Inc. (Industry)
Collaborators: Quintiles, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: TAC101-202
Record Dates: First submitted 2008-05-28; First posted 2008-06-02 (Estimated); Results first posted 2022-02-01 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-08

CONDITIONS: Hepatocellular Carcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — TAC 101

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- TAC-101 (Experimental): Participants with advanced hepatocellular carcinoma who had previously received Sorafenib (as first line therapy) were administered a dose of 20 milligram per day (mg/day) of TAC-101 (as second line treatment) oral tablets within 1 hour post morning meals on Days 1 to 14 followed by a recovery period on Days 15 to 21 in 21-day cycle until disease progression or participant met a treatment discontinuation criterion.
  Interventions: Drug: TAC-101
- Placebo (Placebo Comparator): Participants with advanced hepatocellular carcinoma who had previously received Sorafenib (as first line therapy) were administered a matching placebo for TAC-101 oral tablets within 1 hour post morning meals on Days 1 to 14 followed by a recovery period from on 15 to 21 in 21-day cycle until disease progression or participant met a treatment discontinuation criterion.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: TAC-101 — Participants were randomized to TAC 101 received TAC 101 20 mg (administered as 2 10 mg formulated tablets) PO daily with approximately 240 mL (8 oz) of water under fed conditions (no later than 1 hour after a meal) for 14 days followed by a 7 day recovery period. This cycle was repeated every 21 days.
  Arms: TAC-101
Drug: Placebo — Participants randomized to placebo received 2 placebo tablets (identical in appearance to the TAC 101 tablets) administered PO daily with approximately 240 mL (8 oz) of water under fed conditions (no later than 1 hour after a meal) in a regimen identical to that for TAC 101.
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine whether TAC-101 as a second line therapy for participants who received Sorafenib as first line therapy is effective in slowing tumor activity in patients with advanced hepatocellular carcinoma. The study is also looking at the safety of TAC-101 following treatment with Sorafenib.

DETAILED DESCRIPTION:
Advanced metastatic hepatocellular carcinoma (HCC) is not treatable by surgical approaches or locoregional therapies such as hepatic artery hemoembolization or radiofrequency ablation (RFA) which are effective in controlling localized tumors. Currently marketed systemic chemotherapy agents, with the exception of sorafenib, provide marginal benefit. Despite the demonstrated survival benefit from sorafenib, it is still imperative to improve to the effectiveness of systemic therapy in this patient population. Studies of TAC-101, a synthetic retinoid, indicate that although TAC-101 may not induce tumor regression, it appears to have a stabilizing effect, prolonging survival over what was expected historically. This Phase 2, randomized, double-blind, placebo-controlled international, multicenter study is designed to evaluate the efficacy and safety of TAC 101 as second line treatment in patients with advanced HCC following treatment with sorafenib as first-line therapy. Sorafenib has recently been approved as first line treatment for HCC in the EU and the US and is expected to become the standard of care for the first-line treatment of advanced HCC. Aside from best supportive care, there is no second line therapy available for HCC. It is hypothesized that TAC 101 treatment can extend Overall Survival (OS) after discontinuation of sorafenib.

ELIGIBILITY:
Inclusion Criteria:

* Provide written informed consent prior to performance of any study procedures.
* Is at least 18 years of age.
* Have a diagnosis of advanced unresectable histologically confirmed HCC (excluding fibrolamellar carcinoma).
* Have discontinued from first line treatment with sorafenib monotherapy for any reason (ie, tumor disease progression, intolerance) at least 14 days prior to planned randomization but have not received any second line treatment for HCC.
* Have recovered from any significant sorafenib-related treatment toxicities prior to randomization (Grade 1).
* Have at least 1 target lesion that is viable (has vascularization) and can be accurately measured according to RECIST.
* Patients who have received local therapy prior to sorafenib administration (radiation, surgery, hepatic arterial embolization, chemoembolization, RFA, percutaneous ethanol injection [PEI] or cryoablation) are eligible. Local therapy must be completed at least 4 weeks prior to the baseline scan.
* Have ECOG score of 0, 1, or 2.
* Child-Pugh score <8.
* Have adequate organ function defined as:

  * Platelet count great than 50, less than 109/L;
  * Hemoglobin 8.0 g/dL;
  * Total bilirubin 3 mg/dL;
  * Alanine transaminase (ALT) and aspartate aminotransferase (AST) less than or equal to 5 X ULN;
  * Serum creatinine 1.5 X ULN;
  * PT-international normalized ratio (INR) 2.3 or PT 6 seconds above control
  * Total white blood cell (WBC) count 2.0 109/L
* Is able to take medications orally (eg, no feeding tube).
* Women of childbearing potential must have a negative pregnancy test (urine or serum) prior to randomization and within 2 days prior to starting the study drug. Females must agree to adequate non-estrogenic birth control if conception is possible during the study; and males must agree to adequate birth control during the study and up to 6 months after the discontinuation of study medication.

Exclusion Criteria:

* History of DVT, PE, myocardial infarction (MI), CVA, transitory ischemic attack (TIA), or any other significant TE during the last 3 years.
* Have clinically significant symptoms of hepatic encephalopathy or known brain metastasis.
* Patients who have had clinically significant acute gastrointestinal bleeding as a result of portal vein hypertension within 4 weeks prior to randomization are excluded; however, patients with a history of acute gastrointestinal bleeding that have received appropriate treatment, ie, ligation of varices, are eligible.
* Are receiving therapeutic regimens of anticoagulants, with the exception of prophylaxis care of indwelling venous access devices.
* Have received a liver transplant.
* Are taking prohibited medication.
* Have received a previous systemic therapy (including investigational agents) other than sorafenib (see Inclusion Criterion 4) for treatment of HCC. Patients participating in surveys or observational studies are eligible to participate in this study.
* Have had treatment with any of the following within the specified timeframe prior to randomization:

  * Any sorafenib within the 14 days prior to randomization.
  * Major surgery within the 4 weeks prior to randomization.
  * Any transfusion, treatment with blood component preparation, received. erythropoietin , albumin preparation, and granulocyte colony-stimulating factor (G CSF) within the 2 weeks prior to randomization.
* Has a serious illness or medical condition(s) including, but not limited to the following:

  * Known gastrointestinal disorder, including malabsorption, chronic nausea, vomiting, or diarrhea present to the extent that it might interfere with oral intake and absorption of the study medication.
  * Known human immunodeficiency virus (HIV) or acquired immunodeficiency syndrome (AIDS)-related illness.
  * Previous or concurrent malignancy except for basal cell carcinoma and/or in situ carcinoma of the cervix, or other solid tumor treated curatively and without evidence of recurrence for at least 3 years prior to the study.
  * Uncontrolled metabolic disorders or other nonmalignant organ or systemic diseases or secondary effects of cancer that induce a high medical risk and/or make assessment of survival uncertain.
  * Has active or uncontrolled clinically serious infection excluding chronic hepatitis.
  * Other severe acute or chronic medical or psychiatric condition or laboratory abnormality that may increase the risk associated with study participation or study drug administration, or may interfere with the interpretation of study results, and in the judgment of the Investigator would make the patient inappropriate for entry into this study (eg, active urinary tract infection).
  * Known allergy or hypersensitivity of TAC 101 and any other components used in the TAC 101 tablet.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2008-08-01 (Actual); Primary Completion 2010-05-10 (Actual); Study Completion 2010-05-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Taiho Central, Study Director — Taiho Oncology, Inc. USA
Locations (1):
- I.R.C.C.S. San Matteo University Hospital, Golgi, Pavia, Italy

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 17 study centers worldwide between 01-August-2008 to 10-May-2010.
Pre-assignment Details: The study was stopped after only 52 of the required 220 participants (26 of 110 participants in each treatment group) were randomized. Sponsor terminated the study due to safety concerns and thus, stopped enrollment and study treatment on 06-May-2009, but continued follow-up of all the treated participants for survival till 10 May 2010 and thus, the same was considered as study completion date.
Period: Overall Study
Arm/Group | TAC-101 | Placebo
Started | 26 | 26
Completed | 0 | 0
Not Completed | 26 | 26
Not completed — Adverse Event (AE) | 10 | 3
Not completed — Radiological Disease Progression | 6 | 2
Not completed — Clinical Disease Progression | 1 | 3
Not completed — Investigator Discretion | 3 | 1
Not completed — Sponsor Terminated Study | 6 | 17

BASELINE CHARACTERISTICS:
Population: Baseline analysis included all randomized participants who received any dose of study medication and analyzed by the treatment received.
Groups:
- TAC-101: Participants with advanced hepatocellular carcinoma who had previously received Sorafenib (as first line therapy) were administered a dose of 20 mg/day of TAC-101 (as second line treatment) oral tablets within 1 hour post morning meals on Days 1 to 14 followed by a recovery period on Days 15 to 21 in 21-day cycle until disease progression or participant met a treatment discontinuation criterion.
- Total: Total of all reporting groups
Arm/Group | TAC-101 | Placebo | Total
Number analyzed (Participants) | 26 | 26 | 52
Age, Continuous [Mean (Standard Deviation); unit: years] | 71.1 (6.93) | 68.2 (6.38) | 69.7 (6.75)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 4 | 7
  Male | 23 | 22 | 45
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 23 | 24 | 47
  Black, of African Heritage | 0 | 2 | 2
  Asian | 1 | 0 | 1
  Other: Unspecified | 2 | 0 | 2

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival (OS)
Description: OS was defined as the time from the date of randomization to the date of death. Participants who were still alive were censored at the date last known to be alive (last contact date or last follow-up visit).
Time Frame: From the date of randomization to date of death or up to 1 year post last participant was randomized, whichever was earlier (maximum duration: up to 21.3 months)
Population: Analysis was performed on safety population that included all randomized participants who received at least one dose of double-blind study medication and was summarized by the treatment received.
Measure: Mean (Standard Deviation); unit: months
Arm/Group | TAC-101 | Placebo
Number analyzed (Participants) | 26 | 26
months | 8.23 (5.406) | 8.35 (5.351)

2. Secondary Outcome: Radiologic Progression-free Survival (PFS)
Description: PFS was defined as the time from date of randomization to the date of tumor disease progression (ie, radiological only) or death due to any cause. Participants who were alive at the time of analysis and had no signs of tumor progression had their time of PFS censored at the date of the last tumor assessment, unless they received new antitumor therapy.
Time Frame: From the date of randomization to date of tumor disease progression or death or up to 1 year post last participant was randomized, whichever was earlier (maximum duration: up to 21.3 months)
Population: Analysis was performed on safety population that included all randomized participants who received at least one dose of double-blind study medication and was summarized by the treatment received. Here, 'Overall number of participants analyzed' signifies participants with valid assessment at specified timepoint.
Measure: Mean (Standard Deviation); unit: months
Arm/Group | TAC-101 | Placebo
Number analyzed (Participants) | 21 | 22
months | 4.95 (4.904) | 4.82 (3.647)

3. Secondary Outcome: Time To Progression (TTP)
Description: TTP was defined as time from randomization to the date of tumor progression (radiological only). Participants who were alive with no tumor progression or who died prior to tumor progression had their TTP censored at the date of their last tumor assessment, unless they received new antitumor therapy.
Time Frame: From the date of randomization to date of tumor disease progression or up to 1 year post last participant was randomized, whichever was earlier (maximum duration: up to 21.3 months)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: months
Arm/Group | TAC-101 | Placebo
Number analyzed (Participants) | 21 | 22
months | 4.14 (4.430) | 4.09 (3.146)

4. Secondary Outcome: Number of Participants With Treatment-Emergent Adverse Events (TEAEs) and Treatment-Emergent Serious Adverse Events (TESAEs)
Description: Any untoward medical condition that occurs in a participants while participating in a clinical study and does not necessarily have a causal relationship with the use of the study treatment was considered an AE. A serious AE (SAE) was defined as any untoward medical occurrence that resulted in any of the following outcomes: death, life-threatening, required initial or prolonged in-patient hospitalization, persistent or significant disability/incapacity, congenital anomaly/birth defect, or considered as medically important event. TEAEs were defined as AEs (both serious/non-serious) that occur from the initiation of any study medication administration, and do not necessarily have a causal relationship to the use of the study medication.
Time Frame: From Baseline up to 30 days after the last dose (maximum duration: up to 7.2 months for Placebo and up to 7.9 months for TAC-101)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | TAC-101 | Placebo
Number analyzed (Participants) | 26 | 26
Participants
  TEAE | 26 | 25
  TESAE | 12 | 11

5. Secondary Outcome: Change From Baseline in Plasma Levels of the Tumor Marker Alpha-fetoprotein (AFP)
Description: AFP is a tumor marker for hepatocellular carcinoma and elevations in AFP values could precede clinical deterioration and tumor recurrence in participants. Baseline was defined as the last value obtained within 72 hours prior to study treatment administration on Cycle 1 Day 1.
Time Frame: as for outcome 3
Population: Analysis was performed on safety population that included all randomized participants who received at least 1 dose of double-blind study medication and was summarized by the treatment received. Here, 'Overall number of participants analyzed' signifies participants with valid assessment at specified timepoint.
Measure: Mean (Standard Deviation); unit: nanogram per milliliter (ng/mL)
Arm/Group | TAC-101 | Placebo
Number analyzed (Participants) | 21 | 23
nanogram per milliliter (ng/mL) | 2779.3 (16314.87) | 571.7 (14301.08)

6. Secondary Outcome: Percent Change From Baseline in Plasma Levels of the Tumor Marker Alpha Fetoprotein-L3 (AFP-L3)
Description: AFP-L3 is a tumor marker for hepatocellular carcinoma and elevations in AFP-L3 values could precede clinical deterioration and tumor recurrence in participants. Baseline was defined as the last value obtained within 72 hours prior to study treatment administration on Cycle 1 Day 1.
Time Frame: as for outcome 3
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | TAC-101 | Placebo
Number analyzed (Participants) | 20 | 22
percent change | 2.27 (12.107) | 3.20 (8.129)

7. Secondary Outcome: Maximum Exposure-response Analysis: Maximum Plasma Concentration (Cmax) of TAC-101
Description: Cmax: maximum plasma concentration; Pharmacokinetic (PK) blood samples were collected at 4 hours (± 1 hour), 8 hours (± 1 hour), and 24 hours (± 1 hour) post-dose on Day 1 of treatment Cycle 1. The 24-hour sample was collected prior to dosing on Day 2.
Time Frame: Cycle 1-day 1: 4, 8, and 24 hours after the first dose of study drug
Population: PK population included all participants in safety population participating in this sub-study and treated with active study treatment. Due to limited number of participants with evaluable PK data, no data was collected and analyzed for the conclusion of maximum exposure. Here, 'Overall number of participants analyzed' signifies participants with valid assessment at specified timepoint.
Arm/Group | TAC-101 | Placebo
Number analyzed (Participants) | 0 | 0

8. Secondary Outcome: Overall Exposure-response Analysis: Area Under Curve (AUC0-inf) of TAC-101
Description: AUC(0-inf): Area under the curve from time zero extrapolated to infinity. PK blood samples were collected at 4 hours (± 1 hour), 8 hours (± 1 hour), and 24 hours (± 1 hour) post-dose on Day 1 of treatment Cycle 1. The 24-hour sample was collected prior to dosing on Day 2.
Time Frame: Cycle 1-day 1: 4, 8, and 24 hours after the first dose of study drug
Population: PK population included all participants in safety population participating in this sub-study and treated with active study treatment. Due to limited number of participants with evaluable PK data, no data was collected and analyzed for conclusion of maximum exposure. Here, 'Overall number of participants analyzed' signifies participants with valid assessment at specified timepoint.
Arm/Group | TAC-101 | Placebo
Number analyzed (Participants) | 0 | 0

9. Secondary Outcome: Changes From Baseline in Plasma Insulin-like Growth Factor-2 (IGF-2)
Description: RAR related factors are markers for disease progression in hepatocellular carcinoma participants. In hepatocellular carcinoma participants, IGF-2 is a characteristic biomarkers and its levels are higher in responder cells. The detection of IGF-2 levels showed the efficacy of TAC-101 in IGF-2 influenced malignancy.
Time Frame: From Baseline up to end of study treatment or up to tumor disease progression or up to death or up to 1 year post last participant was randomized, whichever was earlier (maximum duration: up to 21.3 months)
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | TAC-101 | Placebo
Number analyzed (Participants) | 3 | 7
ng/mL | 330.8 (87.82) | 115.6 (181.59)

10. Secondary Outcome: Changes From Baseline in Plasma Transforming Growth Factor-beta (TGFβ2)
Description: TGF-β is responsible for tissue regeneration, cell differentiation, embryonic development, and regulation of the immune system. TGF-β2 levels are higher in non-responder cells hence helps in detection of such cells.
Time Frame: as for outcome 9
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: picograms per milliliter (pg/mL)
Arm/Group | TAC-101 | Placebo
Number analyzed (Participants) | 2 | 7
picograms per milliliter (pg/mL) | -3.51 (4.957) | 0.92 (2.427)

11. Secondary Outcome: Changes From Baseline in Plasma Insulin-like Growth Factor Binding Protein-3 (IGFBP-3)
Description: IGFBP-3 acts as a mediator of antiproliferative signals in hepatocellular carcinoma cells. The inhibition of hepatocellular carcinoma cell proliferation is associated with upregulation of IGFBP-3. Retinoic acid response element (RARE) exists on the promoter region of the IGFBP-3.
Time Frame: as for outcome 9
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | TAC-101 | Placebo
Number analyzed (Participants) | 3 | 7
ng/mL | 370.6 (242.97) | -112.4 (179.64)

12. Secondary Outcome: Changes From Baseline in Plasma Insulin-like Growth Factor Binding Protein-6 (IGFBP-6)
Description: IGFBP-6 has an IGF-2 binding specificity and inhibits growth of a number of IGF-2-dependent cancers. RARE exists on the promoter region of the IGFBP-6.
Time Frame: as for outcome 9
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | TAC-101 | Placebo
Number analyzed (Participants) | 3 | 7
ng/mL | -40.7 (82.08) | -86.9 (72.82)

13. Secondary Outcome: Changes From Baseline in Plasma Lactoferrin
Description: RARE exists on the promoter region of the lactoferrin gene.
Time Frame: as for outcome 9
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | TAC-101 | Placebo
Number analyzed (Participants) | 3 | 6
ng/mL | -133.3 (177.20) | -25.5 (25.83)

14. Secondary Outcome: Changes From Baseline in Plasma Vascular Endothelial Growth Factor-A (VEGF-A)
Description: End of Treatment was defined as "as soon as possible following the last dose of study medication".
Time Frame: as for outcome 9
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | TAC-101 | Placebo
Number analyzed (Participants) | 3 | 7
pg/mL | -29.50 (51.859) | 11.40 (83.141)

15. Secondary Outcome: Number of Participants With Antitumor Activity After Treatment Discontinuation
Description: Antitumor activity after treatment discontinuation in participant was determined by images, computed tomography (CT), and magnetic resonance imaging (MRI). Tumor imaging was done at Baseline any time within 4 weeks prior to the first dose of study treatment on Cycle 1, Day 1 and every 6 weeks (±1 week) during treatment, regardless of a dose delay. If participant discontinued study treatment for a reason other than disease progression (PD), data collected every 6 weeks until PD and following PD, data collected optionally every 6 weeks until death or up to 1 year after the last participant was randomized.
Time Frame: From the date of treatment discontinuation to date of tumor disease progression or death or up to 1 year post last participant was randomized, whichever was earlier (maximum duration: up to 21.3 months)
Population: The data were not collected and analyzed for this outcome measure due to low enrollment of participants.
Arm/Group | TAC-101 | Placebo
Number analyzed (Participants) | 0 | 0

16. Secondary Outcome: Relationship Between Tumor Gene Expression of Messenger Ribonucleic Acid (mRNA) Ratio of Co-activators, Co-repressors and Efficacy Parameters
Description: The assessment of correlative factors was to be conducted on tissue removed prior to the study, if available. Tumor tissue assessments included investigation of the relationship between tumor gene mRNA expression of co-activators and co-repressors and efficacy parameters.
Time Frame: At Baseline (prior to treatment after consenting informed consent form [ICF]) up to last dose of study treatment, assessed every 6 weeks (maximum duration: up to 21.3 months)
Population: The data were not collected and analyzed for this outcome measure due to low enrollment of participants.
Arm/Group | TAC-101 | Placebo
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: From Baseline up to 30 days after the last dose (maximum duration: up to 7.2 months for Placebo and up to 7.9 months for TAC-101)
Description: Analysis was performed on safety population.
Arm/Group | TAC-101 | Placebo
All-Cause Mortality (participants affected / at risk) | 2/26 | 6/26
Serious Adverse Events (participants affected / at risk) | 12/26 | 11/26
Other Adverse Events (participants affected / at risk) | 25/26 | 24/26
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | TAC-101 (N=26) | Placebo (N=26)
Atrial thrombosis (Cardiac disorders) | 2 (2) | 0 (0)
Cardiac arrest (Cardiac disorders) | 0 (0) | 1 (1)
Left ventricular failure (Cardiac disorders) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 2 (2)
Oesophageal varices haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Disease progression (General disorders) | 0 (0) | 1 (1)
Fatigue (General disorders) | 0 (0) | 2 (2)
General physical health deterioration (General disorders) | 0 (0) | 1 (1)
Oedema due to hepatic disease (General disorders) | 1 (1) | 0 (0)
Cytolytic hepatitis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Hepatic failure (Hepatobiliary disorders) | 1 (1) | 1 (1)
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0)
Weight decreased (Investigations) | 0 (0) | 1 (1)
Epilepsy (Nervous system disorders) | 1 (1) | 0 (0)
Hepatic encephalopathy (Nervous system disorders) | 0 (0) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 4 (4) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | TAC-101 (N=26) | Placebo (N=26)
Anaemia (Blood and lymphatic system disorders) | 2 (2) | 2 (2)
Abdominal pain (Gastrointestinal disorders) | 3 (3) | 4 (4)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1) | 2 (2)
Ascites (Gastrointestinal disorders) | 2 (2) | 4 (4)
Constipation (Gastrointestinal disorders) | 0 (0) | 2 (3)
Diarrhoea (Gastrointestinal disorders) | 4 (4) | 5 (5)
Dry mouth (Gastrointestinal disorders) | 2 (2) | 0 (0)
Nausea (Gastrointestinal disorders) | 2 (2) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 3 (3)
Asthenia (General disorders) | 7 (7) | 2 (2)
Fatigue (General disorders) | 6 (8) | 5 (7)
General physical health deterioration (General disorders) | 0 (0) | 2 (2)
Oedema peripheral (General disorders) | 6 (6) | 5 (5)
Performance status decreased (General disorders) | 1 (1) | 3 (3)
Hyperbilirubinaemia (Hepatobiliary disorders) | 2 (2) | 3 (3)
Bronchitis (Infections and infestations) | 1 (1) | 3 (3)
Fall (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Blood bilirubin increased (Investigations) | 2 (2) | 0 (0)
Anorexia (Metabolism and nutrition disorders) | 5 (7) | 2 (2)
Arthralgia (Musculoskeletal and connective tissue disorders) | 5 (5) | 3 (3)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 2 (2)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 4 (4) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 2 (3) | 0 (0)
Dizziness (Nervous system disorders) | 3 (3) | 0 (0)
Headache (Nervous system disorders) | 3 (3) | 0 (0)
Insomnia (Psychiatric disorders) | 0 (0) | 2 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 3 (3)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 2 (3) | 2 (2)
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 3 (4) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 2 (2) | 4 (4)
Rash (Skin and subcutaneous tissue disorders) | 3 (3) | 0 (0)
Hypertension (Vascular disorders) | 2 (4) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 2 (2)

LIMITATIONS AND CAVEATS:
Study was prematurely terminated by Sponsor due to unexpected higher occurrence of thromboembolic events on 06-May-2009. PK & biomarker assessments were optional and explorative,and were not conducted and evaluated due to limited participants count.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other